CLINICAL TRIAL: NCT01357850
Title: A Multi-center, Placebo-controlled Study to Evaluate the Safety of GSK716155 and Its Effects on Myocardial Metabolism, Myocardial Function, and Exercise Capacity in Patients With NYHA Class II/III Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 112670
Record Dates: First submitted 2010-11-11; First posted 2011-05-23 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK716155 (3.75mg) (Experimental): GSK716155 (3.75mg)
  Interventions: Drug: GSK716155
- GSK716155 (15mg) (Experimental): GSK716155 (15mg)
  Interventions: Drug: GSK716155
- GSK716155 (30mg) (Experimental): GSK716155 (30mg)
  Interventions: Drug: GSK716155
- GSK716155-matched placebo (Placebo Comparator): GSK716155-matcued placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK716155 — GSK716155
  Arms: GSK716155 (15mg); GSK716155 (3.75mg); GSK716155 (30mg)
Drug: Placebo — Placebo
  Arms: GSK716155-matched placebo

SUMMARY:
This exploratory proof of concept study will be conducted in patients with stable New York Heart Association (NYHA) Class II-III heart failure. The focus of the efficacy endpoints is to test the hypothesis that GSK716155 administration will increase glucose uptake and utilization in the myocardium, resulting in increased myocardial efficiency and increased exercise capacity. A positive result, defined as either statistically significant effects on one or more of the efficacy endpoints or as an overall signal suggesting a clinically relevant effect on myocardial physiology, would provide evidence for potential progression into further development in a chronic heart failure population.

ELIGIBILITY:
Inclusion Criteria:

* Chronic dilated cardiomyopathy of ischemic or non-ischemic origin
* Clinically stable on optimal therapies for at least 3 months prior to screening/baseline visit.
* Left ventricular ejection fraction greater than or equal to 40% as assessed by any measurement in the previous 24 months.
* NYHA Class II/III heart failure for a minimum of 6 months prior to enrolment
* Male or female between 21 and 75 years of age inclusive, at the time of signing the informed consent. However the optimal age range for this study will be 40 to 65 years of age.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].

Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit ~28 days post-last dose.

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Confirmed QTcB or QTcF < 480 msec; or QTc < 500 msec in subjects with Bundle Branch Block.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Subjects must be able to perform performance/exercise testing

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Active ischemia manifest as a history of myocardial infarction or unstable angina in the past 12 months or a history of coronary revascularization (percutaneous coronary intervention and/or coronary artery bypass grafting) in the past 6 months.

  -. High suspicion of active myocardial ischemia, in the opinion of the treating physician
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* History of drug/alcohol abuse.
* A positive test for HIV antibody.
* Calcitonin > 100 pg./mL
* Triglycerides > 850 mg/dL
* History of significant gastrointestinal surgery, including gastric bypass and banding, antrectomy, Roux-en-Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper gastrointestinal function.
* History of regular alcohol consumption within 6 months of the study defined as:

For UK: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.

For US: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Known allergy or history of sensitivity to albiglutide, any other GLP-1 analogue, , or Baker's yeast.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol (e.g.. related to psychiatric disorder)
* Subject is mentally or legally incapacitated.
* Known diagnosis of diabetes mellitus, fasting glucose >140mg/dL, or HbA1c > 7%.
* Uncorrected thyroid disease manifest as an abnormal thyroid-stimulating hormone (TSH) (outside reference range at screening).
* Other medical problems with life expectancy less than 1yr.
* Other causes of cardiomyopathy or left ventricular dysfunction including:

Uncorrected primary obstructive or regurgitant valvular disease Restrictive cardiomyopathy due to amyloidosis, hemochromatosis, sarcoidosis or other cause Cardiac hypertrophy with wall thickness >1.5cm Alcohol-induced cardiomyopathy Women with heart failure during the 12 months following childbirth. Complex congenital heart disease Anthracycline induced cardiomyopathy

* Subjects with genetic disorders of skeletal muscle (e.g. Duchenne muscular dystrophy)
* Clinically significant pericardial disease.
* Listed as a status 1A or 1B on heart transplant waiting list.
* History of deep vein thrombosis or a known coagulation disorder
* History of pancreatitis
* History of or family history of medullary thyroid carcinoma
* History of or family history of multiple endocrine neoplasia type 2
* History of renal dysfunction with estimated GFR < 40 ml/min at screening
* Resting systolic blood pressure < 85 mmHg or >170 mmHg; or diastolic blood pressure >110 mgHg at screening.
* Inability of the patient to lie flat for a combined total of up to 4 hours to complete imaging assessments.
* No subjects will be enrolled at the single site performing the CMR sub-study who have contraindications to MRI scanning including, but not limited to:

Intracranial aneurysm clips with an appropriate operative conformation History of intra- orbital metal fragments Pacemakers or non-MR compatible heart valves Inner ear implants History of claustrophobia deemed significant by the investigator

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2012-09-18 (Actual); Study Completion 2012-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- United States (12):
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, New York, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
- United Kingdom (3):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lepore JJ, Olson E, Demopoulos L, Haws T, Fang Z, Barbour AM, Fossler M, Davila-Roman VG, Russell SD, Gropler RJ. Effects of the Novel Long-Acting GLP-1 Agonist, Albiglutide, on Cardiac Function, Cardiac Metabolism, and Exercise Capacity in Patients With Chronic Heart Failure and Reduced Ejection Fraction. JACC Heart Fail. 2016 Jul;4(7):559-566. doi: 10.1016/j.jchf.2016.01.008. Epub 2016 Mar 30. PMID 27039125
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 30 day Screening were then randomized to a 13-week Treatment Period, followed by a Follow-up visit 28 days post-treatment. The duration of the study was approximately 20 weeks from Screening to Follow-up. A total of 100 par. were planned, and 82 par. were randomized.
Groups:
- Placebo: Participants received albiglutide matching placebo weekly injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
- Albiglutide 3.75 mg: Participants received albiglutide 3.75 milligrams (mg) weekly injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
- Albiglutide 15 mg: Participants received albiglutide 15 mg weekly injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
- Albiglutide 30 mg: Participants received albiglutide 30 mg weekly injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
Period: Overall Study
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Started | 30 | 12 | 13 | 27
Completed | 29 | 12 | 13 | 27
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Albiglutide 3.75 mg: Participants received albiglutide 3.75 mg weekly injected subcutaneously into the abdomen using a fixed-dose, prefilled, single-use injector pen.
- Total: Total of all reporting groups
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg | Total
Number analyzed (Participants) | 30 | 12 | 13 | 27 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (9.60) | 51.3 (12.44) | 57.2 (11.02) | 58.2 (10.23) | 56.1 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 2 | 7 | 21
  Male | 21 | 9 | 11 | 20 | 61
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 4 | 5 | 4 | 16
  Native Hawaiian Or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 26 | 7 | 8 | 22 | 63
  White - Arabic/North African Heritage | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Myocardial Glucose Utilization as Assessed by [18F]Fluoro-2-deoxy-glucose Positron Emission Tomography (FDG-PET) Imaging
Description: FDG-PET imaging was performed at Baseline and Week 13 to assess myocardial glucose uptake. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on analysis using a mixed effects analysis of variance (ANOVA) model, fitting terms for treatment, visit and interaction of treatment and visit, with participants as random effects.
Time Frame: Baseline and Week 13
Population: Intent-to-Treat (ITT) Population: all randomized participants who received >= 1 dose of study medication and had >= 1 on treatment assessment. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: micromoles per gram per minute
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 10 | 4 | 4 | 11
micromoles per gram per minute | 0.0185 [-0.0158 to 0.0528] | 0.0103 [-0.0440 to 0.0646] | 0.0369 [0.0042 to 0.0695] | 0.0059 [-0.0268 to 0.0386]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 3.75 mg; Test type: Superiority or Other; p = 0.7873, ANOVA; Mean Difference (Final Values) = 0.0119, 95% CI 2-sided [-0.0768 to 0.1005]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 15 mg; Test type: Superiority or Other; p = 0.0499, ANOVA; Mean Difference (Final Values) = 0.0678, 95% CI 2-sided [0.0000 to 0.1356]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 30 mg; Test type: Superiority or Other; p = 0.1666, ANOVA; Mean Difference (Final Values) = 0.0467, 95% CI 2-sided [-0.0204 to 0.1137]

2. Primary Outcome: Change From Baseline in Myocardial Efficiency (Work Performed/Myocardial Oxygen Consumption [MVO2]) Assessed at Rest
Description: MVO2 was estimated by measuring the rate of myocardial clearance of 11C-activity which represents overall myocardial oxidative flux through the TCA cycle. Cardiac work was measured by echocardiography and cardiac efficiency index was calculated as work (by echocardiography) divided by MVO2. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on analysis using a mixed effects ANOVA model, fitting terms for treatment, visit and interaction of treatment and visit, with participants as random effects.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury/liter/minute2
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 10 | 5 | 11 | 11
millimeters of mercury/liter/minute2 | -1051.90 [-3136.43 to 1032.63] | -1070.09 [-3846.14 to 1705.95] | -348.58 [-2278.39 to 1581.23] | -870.64 [-2771.39 to 1030.11]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 3.75 mg; Test type: Superiority or Other; p = 0.9343, ANOVA; Mean Difference (Final Values) = 134.89, 95% CI 2-sided [-3172.05 to 3441.83]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 15 mg; Test type: Superiority or Other; p = 0.3375, ANOVA; Mean Difference (Final Values) = 1278.77, 95% CI 2-sided [-1398.13 to 3955.68]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 30 mg; Test type: Superiority or Other; p = 0.5582, ANOVA; Mean Difference (Final Values) = 772.70, 95% CI 2-sided [-1887.77 to 3433.17]

3. Primary Outcome: Change From Baseline in Peak Oxygen Uptake (Peak VO2) as Assessed by Bicycle Cardiopulmonary Exercise Testing
Description: Peak VO2 was measured at Baseline and Week 13. Participants performed a maximal exercise test limited by dyspnea or fatigue on a cycle ergometer. After a rest period, the workloads were increased in a step fashion by 25 watts every 3 minutes. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on analysis using a mixed effects ANOVA model, fitting terms for treatment, visit and interaction of treatment and visit, with participants as random effects.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliliters per kilogram per minute
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 29 | 12 | 13 | 26
Milliliters per kilogram per minute | -0.63 [-1.53 to 0.27] | 0.05 [-1.35 to 1.45] | 0.51 [-0.84 to 1.85] | 0.88 [-0.07 to 1.83]
Statistical Analysis 1: Comparison: Placebo vs Albiglutide 3.75 mg; Test type: Superiority or Other; p = 0.2256, ANOVA; Median Difference (Final Values) = -2.06, 95% CI 2-sided [-5.43 to 1.30]
Statistical Analysis 2: Comparison: Placebo vs Albiglutide 15 mg; Test type: Superiority or Other; p = 0.5647, ANOVA; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-4.22 to 2.32]
Statistical Analysis 3: Comparison: Placebo vs Albiglutide 30 mg; Test type: Superiority or Other; p = 0.8942, ANOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-2.44 to 2.79]

4. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) as Assessed by Echocardiogram
Description: Echocardiography was performed at Baseline and Week 13 using pulse-wave, continuous-wave, and tissue Doppler. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 28 | 11 | 13 | 27
Percentage | 1.12 (1.06) | 0.99 (2.21) | 1.03 (1.64) | 1.08 (1.08)

5. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Volumes in Systole and Diastole as Assessed by Echocardiogram
Description: Echocardiography was performed at Baseline and Week 13 using pulse-wave, continuous-wave and tissue Doppler. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Milliliters
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 28 | 11 | 13 | 27
Milliliters
  LV end-diastolic volume | 0.9 (4.92) | 1.0 (3.05) | 1.0 (4.37) | 1.0 (5.54)
  LV end-systolic volume | 0.9 (4.05) | 1.0 (3.80) | 1.0 (5.08) | 0.9 (5.11)

6. Secondary Outcome: Change From Baseline in LV and RV Function Assessed by Cardiac Magnetic Resonance (CMR) (LVEF), Myocardial Strain Assessed by Myocardial Tagging Indices
Description: Non-contrast CMR to assess left ventricular (LV) and right ventricular (RV) ejection fraction, volume, mass, and strain was performed following a period of rest after exercise testing at Baseline and after the Week 13 treatment phase. A 3Tesla magnetic resonance imagine (MRI) examination was performed including sequences for evaluation of LV structure and function. Only those participants available at the specified time points were analyzed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: CMR Substudy Population: all randomized participants who participated in the CMR substudy and had valid Baseline and/or Week 13 assessments for >= 1 one of the imaging parameters of LV and RV function assessed by CMR (LVEF, LV and RV volumes in systole and diastole, LV mass), myocardial strain assessed by myocardial tagging indices.
Measure: Geometric Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 5 | 1 | 2 | 7
Percentage | 1.17 (1.64) | 1.14 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the mean and standard error cannot be calculated. | 1.09 (4.0) | 1.09 (1.90)

7. Secondary Outcome: Change From Baseline in LV and RV Function Assessed by CMR (LV and RV Volumes in Systole and Diastole), Myocardial Strain Assessed by Myocardial Tagging Indices
Description: Non-contrast CMR to assess LV and RV ejection fraction, volume, mass, and strain was performed following a period of rest after exercise testing at Baseline and after the Week 13 treatment phase. A 3Tesla magnetic resonance imagine (MRI) examination was performed including sequences for evaluation of LV structure and function. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: CMR Substudy Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Milliliters
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 5 | 1 | 2 | 7
Milliliters
  LV end-diastolic volume | 0.99 (11.08) | 1.02 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the mean and standard error cannot be calculated. | 0.96 (12.50) | 0.95 (11.79)
  LV end-systolic volume | 0.90 (7.80) | 0.89 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the mean and standard error cannot be calculated. | 0.94 (3.00) | 0.89 (9.42)

8. Secondary Outcome: Change From Baseline in LV and RV Function Assessed by CMR (LV Mass), Myocardial Strain Assessed by Myocardial Tagging Indices
Description: Non-contrast CMR to assess left/right ventricular ejection fraction, volume, mass, and strain was performed following a period of rest after exercise testing at Baseline and after the Week 13 treatment phase. A 3Tesla magnetic resonance imagine (MRI) examination was performed including sequences for evaluation of LV structure and function. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: CMR Substudy Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Grams
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 5 | 1 | 2 | 7
Grams | 0.96 (7.99) | 1.04 (NA) — Only one participant was analyzed in this treatment arm at this time point; therefore the mean and standard error cannot be calculated. | 1.08 (1.50) | 0.97 (10.65)

9. Secondary Outcome: Change From Baseline in Cardiac Energetics (PCr/ATP) Measured by 31P Magnetic Resonance Spectroscopy (MRS)
Description: Participants underwent a CMR scan performed on a 3 Tesla MR system at Baseline and Week 13 to assess cardiac mass, volumes (global function and dilatation), strain and torsion, cardiac and liver lipid content and cardiac energy metabolism. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: Magnetic Resonance Substudy Population (MRS): all randomized participants who participated in the MRS substudy and had valid Baseline and/or Week 13 assessments for either PCr/ATP via 31P MRS. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Albiglutide 30 mg
Number analyzed (Participants) | 5 | 6
ratio | 0.33 [-0.29 to 0.94] | 0.11 [-0.45 to 0.67]

10. Secondary Outcome: Change From Baseline in Cardiac and Liver Fat by Proton Spectroscopy (1H MRS)
Description: Change in Baseline in cardiac and liver fat by proton spectroscopy was planned at Baseline and Week 13. The protocol allowed for sites to perform all or only efficacy assessments, depending on site designation, capability and feasibility. No sites that enrolled participants into this study were able to perform this outcome measure.
Time Frame: Baseline and Week 13
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Exercise Capacity Assessed by 6-minute Walk Test
Description: The six minute walk test was performed at Baseline and Week 13. All participantss were given standardized instructions and the distance walked was measured. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Meters
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 28 | 12 | 13 | 27
Meters | 1.03 [0.98 to 1.07] | 1.10 [0.96 to 1.25] | 1.14 [1.00 to 1.30] | 1.05 [1.00 to 1.10]

12. Secondary Outcome: Change From Baseline in Serum N-terminal Fragment Brain Natriuretic Peptide (NT-BNP) Level
Description: Baseline is defined as the last available assessment on or prior to the first dose of study medication. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Change from Baseline at Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: Nanogram per liter
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 28 | 12 | 12 | 25
Nanogram per liter | 0.90 (10.43) | 0.90 (34.20) | 0.70 (31.50) | 0.90 (25.73)

13. Secondary Outcome: Change From Baseline in Plasma Levels of Glucose, and Free Fatty Acids (FFA)
Description: Blood samples for biomarker analysis of fasting levels of glucose and FFA were collected at Weeks 1, 7 and 13; glucose was also collected at Weeks 2, 4, 6, 8, 10, and 12. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X in the category titles). Different participants may have been analyzed for different parameters at different time points, so the overall number of participants analyzed reflects everyone in the ITT population.
Measure: Geometric Mean (Standard Error); unit: Millimole per liter (mmol/L)
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 30 | 12 | 13 | 27
Millimole per liter (mmol/L)
  FFA (n=24, 10, 12, 22) | 0.81 (0.03) | 0.90 (0.05) | 0.74 (0.04) | 0.87 (0.05)
  Glucose (n=29, 12, 13, 27) | 1.01 (0.14) | 0.91 (0.27) | 1.00 (0.16) | 1.00 (0.17)

14. Secondary Outcome: Change From Baseline in Plasma Levels of Insulin
Description: Blood samples for biomarker analysis of fasting levels of insulin were collected at Weeks 1, 7 and 13. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Standard Error); unit: picomole per liter (pmol/L)
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 28 | 12 | 13 | 26
picomole per liter (pmol/L) | 0.9 (18.08) | 0.7 (30.49) | 1.0 (15.41) | 1.2 (15.56)

15. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the Minnesota Living With Heart Failure Questionnaire
Description: Minnesota living with heart failure questionnaire (MLHFQ) is a validated instrument to measure participant-reported quality of life at Baseline and Week 13. For each of 21 items, participants rated the effects of heart failure and its treatment on physical, socioeconomic and psychological aspects of their life. To measure the effects of symptoms, functional limitations, psychological distress on an individual's quality of life, the MLHF questionnaire asks each participant to indicate their response using a 6-point scale (ranging from 0 to 5, 0=no, 1=very little, and 5=very much). The min and max scores can range from 0 to 105. The likert scale measures the effect of heart failure and treatments for heart failure on an individual's ability to live as they want. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 13
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 29 | 12 | 13 | 27
Scores on a scale | 0.8 [0.6 to 1.0] | 0.7 [0.4 to 1.2] | 0.7 [0.5 to 1.0] | 0.7 [0.5 to 0.9]

16. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Please refer to the AE/SAE section for further details.
Time Frame: Baseline and Week 13
Population: All Subject Population: all randomized participants who received >= 1 dose of study medication. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 30 | 12 | 13 | 27
Participants
  Any AE | 25 | 12 | 12 | 20
  Any SAEs | 4 | 2 | 2 | 0

17. Secondary Outcome: Number of Participants With Adverse Events by the Indicated Severity
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect. Severity categories: Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities;Moderate: an event that was sufficiently discomforting to interfere with normal everyday activities; Severe: an event that prevents normal everyday activities.
Time Frame: Baseline and Week 13
Population: All Subjects Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Number analyzed (Participants) | 30 | 12 | 13 | 27
Participants
  Mild | 10 | 6 | 4 | 12
  Moderate | 13 | 4 | 6 | 6
  Severe | 2 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs collected from the start of study medication and within 30 days after the end of study medication (Week 13) are reported.
Description: AEs and non-serious AEs are reported for members of the All subjects Population, comprised of all participants randomized to treatment, who have taken at least one dose of study medication.
Arm/Group | Placebo | Albiglutide 3.75 mg | Albiglutide 15 mg | Albiglutide 30 mg
Serious Adverse Events (participants affected / at risk) | 4/30 | 2/12 | 2/13 | 0/27
Other Adverse Events (participants affected / at risk) | 22/30 | 11/12 | 11/13 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Albiglutide 3.75 mg (N=12) | Albiglutide 15 mg (N=13) | Albiglutide 30 mg (N=27)
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Device Malfunction (General disorders) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Albiglutide 3.75 mg (N=12) | Albiglutide 15 mg (N=13) | Albiglutide 30 mg (N=27)
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3 | 4
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 1
Ear infection (Infections and infestations) | 0 | 2 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 2
Injection site pruritus (General disorders) | 1 | 1 | 0 | 1
Injection site haematoma (General disorders) | 1 | 2 | 2 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 0
Implant site pain (General disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 3
Lipase increased (Investigations) | 0 | 0 | 0 | 3
Blood urea increased (Investigations) | 1 | 1 | 0 | 2
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Gout (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Acne cystic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.